CLINICAL TRIAL: NCT01246687
Title: Dietary Intervention Among Patients With Type 2 Diabetes Mellitus: An e-Approach
Brief Title: Web-based Dietary Intervention for Diabetic Patients
Acronym: myDIDeA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Amutha Ramadas, Ms, Monash University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MED2009-CM(SG)-004-QKF
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus, Type 2; Intervention Studies; Behavior
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Behavior

ARMS (2):
- e-Intervention group (Experimental): Receive stage-specific dietary intervention via the website & standard care at the outpatient clinic.
  Interventions: Behavioral: e-Intervention
- Control group (No Intervention): Continue with the standard diabetes care at the outpatient clinic without getting access to the web-based intervention.

INTERVENTIONS:
Behavioral: e-Intervention — Dietary educational programme developed using Transtheoretical Model of Change and delivered via a website specific for Type 2 Diabetes patients.
  Arms: e-Intervention group

SUMMARY:
The Internet holds promise for a wide-scale promotion of dietary and lifestyle behavioural change. Website-delivered interventions have a potentially broad population reach as it is available 24 hours, and could be hosted by both government and non-governmental agencies. To date, there is no published study focused on dietary behaviour change in adults with Type 2 Diabetes Mellitus (T2DM) via a website-based system.

myDIDeA was a 12-months two-armed randomised controlled trial conducted in three tertiary public hospitals in Klang Valley, Malaysia. The primary outcome was the Dietary Knowledge, Attitude and Behaviour (DKAB) score, while the secondary outcomes included the food intake, anthropometry measurements, blood pressure and resting heart rate, blood biomarkers and the Dietary Stages of Change (DSOC) score.

DETAILED DESCRIPTION:
The study was designed according to the recommendations of the CONSORT statement for randomised trials of non-pharmacologic treatment. The study commenced in November 2009 after obtaining the ethical approvals from relevant authorities, and the trial has been registered with Clinicaltrials.gov (NCT01246687). After being screened for eligibility, 128 patients with Type 2 Diabetes Mellitus (T2DM) from the outpatient clinics at these hospitals were recruited into the study with informed consent. After the baseline data collection, the participants were randomised into the e-intervention (n=66) or the control (n=62) group. The e-intervention group received an intensive six-month dietary intervention through the study website, which was developed based on various established guidelines and recommendations but personalised according to the participants' DSOC, in addition to the usual standard treatment at the outpatient clinics. In contrast, the control group received the usual standard treatment given to patients with T2DM, and did not receive the website login information, or any reinforcement via e-mail or SMS. Data were collected at baseline, six months post-intervention and at 12 months follow-up. A structured and pre-tested questionnaire was used for this purpose. The anthropometry measurements, blood pressure and resting heart rate were measured at data collection. Details on the blood biomarkers were obtained from the hospital medical records. The statistical analysis revealed that myDIDeA was successful in improving overall DKAB score by improving the diabetes-related dietary knowledge and attitude of the participants. Besides, the intervention programme also have successfully improved the DSOC score of the intervention group, suggesting the participants were indeed making small but significant progress in changing their dietary behaviour. Improvement in the diet quality (improvement in vegetable intake and reduction in carbohydrate and protein intake), glycaemic control and total cholesterol have added credibility to this web-delivered intervention. The process evaluation of the study website revealed that on the average each participant logged in the website once a week and spent 11 minutes at the website per visit. The usability (facilitating conditions) scored the highest, while the acceptability (anxiety) scored the lowest.

ELIGIBILITY:
Inclusion Criteria:

* Mentally sound men and women who are > 18 years old.
* Literate with a fair command of English and/or Malay languages.
* Have access to the Internet at home, work or public place.
* Willing to access the web portal at least once every fortnight.
* Have been confirmed to have HbA1c of >7%.
* KAB score < 50% at baseline.

Exclusion Criteria:

* Pregnant, lactating or intend to become pregnant during the study period.
* Diagnosed with Type 1 Diabetes Mellitus (T1DM) or Gestational Diabetes Mellitus (GDM)
* Weighing not more than 150% of the desired weight for height.
* Any pre-existing condition compromising the quality of life or ability to participate according to protocol.
* Have severe complications (chronic heart disease, cerebrovascular disease, diagnosed HIV/AIDS, cancer, emphysema, chronic liver or kidney disease) that would affect the subjects' ability to follow the tailored advice.
* Enrolled in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Dietary KAB Score at 6 months | Baseline & 6 months
  Dietary Knowledge, Attitude & Behaviour Score - assessed using 36-item questionnaire.
Change from Baseline in Dietary KAB Score at 12 months | Baseline & 12 months
  Dietary Knowledge, Attitude & Behaviour Score - assessed using 36-item questionnaire.

SECONDARY OUTCOMES:
Change from Baseline in anthropometric measurements at 6 months | Baseline & 6 months
  BMI, body fat percentage, waist circumference
Change from Baseline in anthropometric measurements at 12 months | Baseline & 12 months
  BMI, body fat percentage, waist circumference
Change from Baseline in dietary practices at 6 months | Baseline & 6 months
  Nutrient intake, dietary GI, supplement intake, food preparation & eating out habit
Change from Baseline in dietary practices at 12 months | Baseline & 12 months
  Nutrient intake, dietary GI, supplement intake, food preparation & eating out habit
Change from Baseline in blood biomarkers at 6 months | Baseline & 6 months
  HbA1c, fasting plasma glucose, lipid profile (data to be obtained from the medical records)
Change from Baseline in blood biomarkers at 12 months | Baseline & 12 months
  HbA1c, fasting plasma glucose, lipid profile (data to be obtained from the medical records)

CONTACTS AND LOCATIONS:
Overall Officials: Kia Fatt Quek, PhD, Principal Investigator — Monash University (Sunway Campus)
Locations (3):
- Malaysia (3):
  - Hospital Putrajaya, Putrajaya, Putrajaya
  - Hospital Selayang, Batu Caves, Selangor
  - Hospital Serdang, Kajang, Selangor

REFERENCES:
- [Derived] Ramadas A, Chan CKY, Oldenburg B, Hussein Z, Quek KF. Randomised-controlled trial of a web-based dietary intervention for patients with type 2 diabetes: changes in health cognitions and glycemic control. BMC Public Health. 2018 Jun 8;18(1):716. doi: 10.1186/s12889-018-5640-1. PMID 29884161
- [Derived] Ramadas A, Quek KF, Chan CK, Oldenburg B, Hussein Z. Randomised-controlled trial of a web-based dietary intervention for patients with type 2 diabetes mellitus: study protocol of myDIDeA. BMC Public Health. 2011 May 21;11:359. doi: 10.1186/1471-2458-11-359. PMID 21599990